CLINICAL TRIAL: NCT00893828
Title: Monitoring Pulmonary Artery Pressure by Implanted Device Responding to Ultrasonic Signal
Brief Title: Monitoring Pulmonary Artery Pressure by Implantable Device Responding to Ultrasonic Signal (PAPIRUS III)
Acronym: PAPIRUSIII
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Rev. B, 29-Sep-08
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The PAPIRUS III study will continue to follow patients initially enrolled in PAPIRUS II. Pressure readings from the investigational device will continue to be collected and will be correlated to physiological changes during activities of daily living and protocol defined tests.

DETAILED DESCRIPTION:
This is a small clinical trial to determine the feasibility of a device & to test prototype device, where the primary outcome measure relates to feasibility and not to health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been enrolled in the PAPIRUS II Study and has a RemonCHF pressure sensor implanted
* Patient is willing and able to provide informed consent, participate in the Safety Follow-up Program and/or in the required tests associated with the clinical investigation (Core Study Program) at an approved clinical investigational center and at the intervals defined by the Clinical Investigational Plan.

Exclusion Criteria:

* Patient enrolled in PAPIRUS II but not implanted with a RemonCHF Pressure Sensor
* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study (with the exception of the PAPIRUS II Study). Each instance would be brought to the sponsor to determine eligibility.
* Age < 18 years
* Women of childbearing potential who are, or might be, pregnant at the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously implanted with a RemonCHF device
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Continue detailed data collection of pressure readings from patients implanted with a RemonCHF device. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Uta C Hoppe, Prof. Dr., Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided